CLINICAL TRIAL: NCT05567185
Title: A Phase 1 Study to Evaluate the Tolerability, Safety, and Pharmacokinetics of TAR-210 in Japanese Participants With Bladder Cancer and Selected FGFR Mutations or Fusions
Brief Title: A Study of Erdafitinib Intravesical Delivery System in Japanese Participants With Bladder Cancer
Acronym: TAR-210
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109248; 42756493BLC1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder Neoplasms; Receptors, Fibroblast Growth Factor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Acrocephalosyndactylia | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation: Erdafinitib Intravesical Delivery System (Experimental): Participants with bladder cancer and fibroblast growth factor receptor (FGFR) mutations or fusions will receive erdafitinib intravesical delivery system and study will evaluate 2 dose levels of erdafitinib. Participants with a complete response (CR) may continue to receive treatment up to a duration of 1 year as long as there is no disease recurrence or progression, intolerable toxicity or withdrawal of consent.
  Interventions: Drug: Erdafitinib Intravesical Delivery System

INTERVENTIONS:
Drug: Erdafitinib Intravesical Delivery System — Erdafitinib intravesical delivery system will be administered.
  Other Names: JNJ-42756493

SUMMARY:
The purpose of the study is to determine the tolerability of erdafitinib intravesical delivery system (TAR-210) in Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-muscle-invasive urothelial carcinoma of the bladder
* All visible tumors must be completely resected prior to the start of study treatment and documented on screening cystoscopy
* Confirmed recurrence of non-muscle invasive bladder cancer (NMIBC) after prior therapy that meet either one: a. Recurrence of high-risk NMIBC (high-grade Ta or any-grade T1) within 12 months after adequate Bacillus Calmette-Guerin (BCG), or any-grade T1 within 3 months after 1st induction course, refusing or ineligible for radical cystectomy (RC). b. Recurrence of intermediate- or high-risk NMIBC (any-grade Ta/T1) after prior BCG regardless of the timing of recurrence, refusing or ineligible for RC and considering no other effective treatment options. c. Recurrence of intermediate-risk NMIBC (low grade Ta) after intravesical chemotherapy including maintenance therapy following a single dose after operation, no other effective intravesical chemotherapy is available and refusing BCG treatment
* At least 1 of the study protocol defined activating fibroblast growth factor receptors (FGFR) mutation or fusion, as determined by local or central testing using either tumor tissue or urine sample collected prior to trans urethral resection of bladder tumour (TURBT)
* Eastern Cooperative Oncology Group (ECOG) performance status score of less than or equal to (<=) 2

Exclusion Criteria:

* Histologically confirmed muscle-invasive (T2 or higher stage) urothelial carcinoma of the bladder.
* Prior treatment with an fibroblast growth factor receptor (FGFR) inhibitor
* Presence of any bladder or urethral anatomic feature that in the opinion of the investigator may prevent the safe placement, indwelling use, or removal of erdafitinib intravesical delivery system
* Participants with active bladder stones or history of bladder stones less than [< 6] months prior to the start of study treatment
* Participants have concurrent or second malignancy other than the disease which natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s); -Bladder post-void residual volume (PVR) >350 mL after second voided urine, -Current central serous retinopathy or retinal pigment epithelial detachment of any-grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2027-09-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events related to erdafitinib intravesical delivery system and are defined as any of the following: high grade non-hematologic toxicity or hematologic toxicity.

SECONDARY OUTCOMES:
Plasma Concentration of Erdafitinib | Up to 180 days
  Plasma concentration of erdafitinib will be reported.
Urine Concentration of Erdafitinib | Up to 180 days
  Urine concentration of erdafitinib will be reported.
Number of Participants with Adverse Events (AEs) | Up to 3 years 10 months
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with AEs by Severity | Up to 3 years 10 months
  Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (4):
- Japan (4):
  - St Marianna University Hospital, Kanagawa
  - Osaka International Cancer Institute, Osaka
  - Toyama University Hospital, Toyama
  - University of Tsukuba Hospital, Tsukuba

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency